CLINICAL TRIAL: NCT01882803
Title: A Phase 2 Study of Duvelisib in Subjects With Refractory Indolent Non-Hodgkin Lymphoma
Brief Title: A Study of Duvelisib in Participants With Refractory Indolent Non-Hodgkin Lymphoma
Acronym: DYNAMO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-145-06; 2013-004008-20 (EudraCT Number)
Record Dates: First submitted 2013-05-31; First posted 2013-06-20 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Indolent Non-Hodgkin Lymphoma
Keywords: PI3K Inhibitor
MeSH Terms: interventions — duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Duvelisib (Experimental)
  Interventions: Drug: Duvelisib

INTERVENTIONS:
Drug: Duvelisib — Phosphoinositide-3-kinase (PI3K) inhibitor
  Other Names: Copiktra; IPI-145

SUMMARY:
This was a Phase 2 clinical trial to evaluate the safety and efficacy of duvelisib as a monotherapy in participants with indolent non-Hodgkin lymphoma (iNHL) (follicular lymphoma [FL], marginal zone lymphoma, or small lymphocytic lymphoma) that was refractory to rituximab and to either chemotherapy or radioimmunotherapy (RIT).

DETAILED DESCRIPTION:
This was an open-label, single-arm safety and efficacy study of duvelisib administered orally to participants who had been diagnosed with iNHL whose disease was refractory to rituximab and to either chemotherapy or RIT.

Approximately 120 participants received 25 milligrams of duvelisib twice daily over the course of 28-day treatment cycles for up to 13 cycles.

After completing 13 treatment cycles of duvelisib, participants continued to receive additional cycles of duvelisib until disease progression or unacceptable toxicity. However, to receive additional cycles of duvelisib beyond 13 cycles, participants must have had evidence of response (complete response [CR] or partial response [PR]) or stable disease according to the International Working Group criteria by the end of Cycle 13.

ELIGIBILITY:
Inclusion Criteria:

* Participants who had been diagnosed with iNHL that had progressed.
* Participants must have exhibited lack of CR or progressive disease (PR) or progression within 6 months after the last dose of a chemotherapy induction regimen or RIT.
* Participants must have had rituximab-refractory disease, defined as lack of CR or PR or PD within 6 months of last dose.
* Measurable disease with a lymph node or tumor mass ≥1.5 centimeters in at least one dimension by computed tomography (CT), positron emission tomography/CT or magnetic resonance imaging.
* Adequate renal and hepatic function.

Exclusion Criteria:

* Candidate for potentially curative therapies in the opinion of the investigator.
* Previous treatment with a PI3K inhibitor or Bruton's tyrosine kinase inhibitor.
* Prior history of allogeneic hematopoietic stem cell transplant.
* Prior chemotherapy, cancer immunosuppressive therapy, or other investigational agents within 4 weeks before first dose of study drug.
* Grade 3B FL and/or clinical evidence of transformation to a more aggressive subtype of lymphoma.
* Symptomatic central nervous system NHL.
* Ongoing systemic bacterial, fungal, or viral infections at the time of initiation of study treatment.
* Prior, current, or chronic hepatitis B or hepatitis C infection, positive result for hepatitis C virus antibodies, hepatitis B surface antigen, or hepatitis B core antibodies.
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2013-06-17 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (63):
- United States (23):
  - Los Angeles, California
  - Whittier, California
  - Denver, Colorado
  - Fort Myers, Florida
  - St. Petersburg, Florida
  - Tallahassee, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - St Louis, Missouri
  - Howell Township, New Jersey
  - Morristown, New Jersey
  - New York, New York
  - Rockville Centre, New York
  - Canton, Ohio
  - Lawton, Oklahoma
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Lynchburg, Virginia
- Belarus (4):
  - Lyasny, Minsk Oblast
  - Brest
  - Minsk
  - Vitebsk
- Belgium (2):
  - Ghent
  - Kortrijk
- Sofia, Bulgaria
- Canada (3):
  - Toronto, Ontario
  - Gatineau, Quebec
  - Montreal, Quebec
- Czechia (2):
  - Brno
  - Ostrava-Poruba
- France (5):
  - Angers
  - Bordeaux
  - Clermont-Ferrand
  - Marseille
  - Pierre-Bénite
- Tbilisi, Georgia
- Hungary (2):
  - Budapest
  - Debrecen
- Italy (12):
  - Bologna
  - Brescia
  - Busto Arsizio
  - Genova
  - Meldola
  - Milan
  - Modena
  - Orbassano
  - Parma
  - Ravenna
  - Rimini
  - Varese
- Spain (3):
  - Barcelona
  - Madrid
  - Salamanca
- United Kingdom (5):
  - Cardiff
  - Chelsea
  - Liverpool
  - London
  - Sutton

REFERENCES:
- [Derived] Flinn IW, Miller CB, Ardeshna KM, Tetreault S, Assouline SE, Mayer J, Merli M, Lunin SD, Pettitt AR, Nagy Z, Tournilhac O, Abou-Nassar KE, Crump M, Jacobsen ED, de Vos S, Kelly VM, Shi W, Steelman L, Le N, Weaver DT, Lustgarten S, Wagner-Johnston ND, Zinzani PL. DYNAMO: A Phase II Study of Duvelisib (IPI-145) in Patients With Refractory Indolent Non-Hodgkin Lymphoma. J Clin Oncol. 2019 Apr 10;37(11):912-922. doi: 10.1200/JCO.18.00915. Epub 2019 Feb 11. PMID 30742566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter, multinational study enrolled participants at 56 medical clinics across 12 countries.
Groups:
- Duvelisib: Participants received a dose of 25 milligrams (mg) duvelisib twice daily (BID) over the course of 28-day treatment cycles until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Duvelisib
Started | 129
Received at Least 1 Dose of Study Drug | 129 (Participant received treatment in 28-day cycles until disease progression or unacceptable toxicity.)
Completed | 0
Not Completed | 129
Not completed — Disease Progression | 1
Not completed — Withdrawal by Subject | 9
Not completed — Death | 68
Not completed — Physician Decision | 3
Not completed — Lost to Follow-up | 3
Not completed — Follow-up Completed | 39
Not completed — Study Terminated by the Sponsor | 6

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of duvelisib.
Groups:
- Duvelisib: Participants received a dose of 25 mg duvelisib BID over the course of 28-day treatment cycles until disease progression or unacceptable toxicity.
Arm/Group | Duvelisib
Number analyzed (Participants) | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 118
  Unknown or Not Reported | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1
  Asian | 1
  Black or African American | 6
  Native Hawaiian or other Pacific Islander | 0
  White | 116
  Other | 1
  Unknown | 2
  Missing | 2
Region of Enrollment [Number; unit: participants]
  Hungary | 7
  United States | 46
  Czechia | 9
  United Kingdom | 11
  Belarus | 10
  Spain | 2
  Canada | 9
  Belgium | 2
  Italy | 21
  Georgia | 1
  France | 6
  Bulgaria | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR, defined as the total percentage of participants who had a best overall response of either complete response (CR) or partial response (PR), was evaluated locally (investigator's assessment) according to the revised IWG Response Criteria for Malignant Lymphoma. ORR is reported with a 2-sided 95% exact confidence interval.
Time Frame: Every 8-16 weeks while on treatment with duvelisib for up to 72 months
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of duvelisib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Duvelisib
Number analyzed (Participants) | 129
percentage of participants | 59.7 [50.7 to 68.2]
Statistical Analysis 1: Comparison: Duvelisib; ORR was tested against the null (≤30%) by 1-sided exact binomial test at 0.025 level; Test type: Other; p <= 0.0001, Exact Binomial Test — '<=' represents '≤'; The p-value was calculated by 1-sided exact binomial test with the null hypothesis that ORR ≤30%

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A TEAE was defined as any adverse event that emerged or worsened in the period from the first dose of study treatment to 30 days after the last dose of study treatment. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Every 2-8 weeks for up to 73 months
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of duvelisib.
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib
Number analyzed (Participants) | 129
Participants | 128

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR, defined as the time from the first documentation of response to either progressive disease (PD) or death due to any cause, was evaluated locally (investigator's assessment) according to the revised IWG Response Criteria for Malignant Lymphoma.
Time Frame: Every 8-16 weeks for up to 72 months
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of duvelisib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Duvelisib
Number analyzed (Participants) | 129
months | 10.16 [8.78 to 13.61]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS, defined as the time from the first dose of study treatment to the first documentation of either Investigator-assessed PD or death resulting from any cause, was evaluated locally (investigator's assessment) according to the revised IWG Response Criteria for Malignant Lymphoma.
Time Frame: Every 8-16 weeks for up to 72 months
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of duvelisib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Duvelisib
Number analyzed (Participants) | 129
months | 9.57 [8.35 to 11.70]

5. Secondary Outcome: Overall Survival (OS)
Description: OS, defined as the time from the first dose of study treatment to the date of death, was evaluated locally (investigator's assessment) according to the revised IWG Response Criteria for Malignant Lymphoma.
Time Frame: Every 16 weeks for up to 72 months
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of duvelisib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Duvelisib
Number analyzed (Participants) | 129
months | 28.96 [21.37 to 37.02]

6. Secondary Outcome: Plasma Concentration of Duvelisib and IPI-656
Description: The serum concentration of duvelisib and its main metabolite, IPI-656, are reported for Day 15 of Cycle 1 (C1D15) and Day 1 of Cycle 2 (C2D1) and Day 1 of Cycle 3 (C3D1). Results are reported in nanograms/milliliter (ng/mL).
Time Frame: Every 4 weeks for 12 weeks (C1D15: predose, 1 and 4 hours post dose; C2D1 and C3D1: anytime during study visit)
Population: Pharmacokinetics (PK) Set: all participants who received at least 1 dose of duvelisib and with at least 1 adequate post-baseline blood sample.
Measure: Median (Full Range); unit: ng/mL
Groups:
- IPI-656: Participants who received at least 1 dose of duvelisib and with at least 1 adequate post-baseline blood sample for measuring concentrations of the main duvelisib metabolite, IPI-656.
Arm/Group | Duvelisib | IPI-656
Number analyzed (Participants) | 129 | 129
ng/mL
  C1D15 Predose: number analyzed (Participants) | 117 | 117
  C1D15 Predose | 414 [19 to 4590] | 648 [116 to 6010]
  C1D15 1 hour post dose: number analyzed (Participants) | 118 | 118
  C1D15 1 hour post dose | 1175 [206 to 6820] | 641 [160 to 5920]
  C1D15 4 hours post dose: number analyzed (Participants) | 129 | 118
  C1D15 4 hours post dose | 852 [233 to 5170] | 714 [230 to 6020]
  C2D1: number analyzed (Participants) | 129 | 117
  C2D1 | 631 [NA to 4180] — <lower limit of quantification | 704 [NA to 10200] — <lower limit of quantification
  C3D1: number analyzed (Participants) | 110 | 110
  C3D1 | 696 [NA to 3540] — <lower limit of quantification | 664 [NA to 6850] — <lower limit of quantification

7. Secondary Outcome: Time to Response (TTR)
Description: TTR, defined as the time from the first dose of study treatment to the first documentation of response, was evaluated by an independent, third-party panel of radiologists and oncologists (Independent Review Committee [IRC]) according to the revised IWG Response Criteria for Malignant Lymphoma.
Time Frame: First dose to first documentation of complete or partial response (up to 6 months)
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of duvelisib and who were considered responders (CR or PR) per IRC.
Measure: Median (Inter-Quartile Range); unit: month
Arm/Group | Duvelisib
Number analyzed (Participants) | 59
month | 1.87 [1.71 to 3.65]

ADVERSE EVENTS:
Time Frame: 73 months
Arm/Group | Duvelisib
All-Cause Mortality (participants affected / at risk) | 68/129
Serious Adverse Events (participants affected / at risk) | 83/129
Other Adverse Events (participants affected / at risk) | 122/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Duvelisib (N=129)
Febrile neutropenia (Blood and lymphatic system disorders) | 9
Pancytopenia (Blood and lymphatic system disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 10
Colitis (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal mass (Gastrointestinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 9
Pyrexia (General disorders) | 4
Fatigue (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 7
Bronchopneumonia (Infections and infestations) | 4
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Clostridium difficile colitis (Infections and infestations) | 1
Cystitis pseudomonal (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infective myositis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Klebsiella sepsis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Neutropenic sepsis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 2
Oropharyngeal candidiasis (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1
Pneumonia pseudomonas aeruginosa (Infections and infestations) | 2
Pseudomembranous colitis (Infections and infestations) | 1
Pseudomonal bacteraemia (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Scrotal infection (Infections and infestations) | 1/88 — This adverse event only affected male participants.
Sepsis (Infections and infestations) | 1
Sepsis syndrome (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Vulval cellulitis (Infections and infestations) | 1/41 — This adverse event only affected female participants.
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 4
Renal failure (Renal and urinary disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Peripheral embolism (Vascular disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Glaucoma (Eye disorders) | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 2
Bronchitis (Infections and infestations) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Campylobacter infection (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Pneumonia moraxella (Infections and infestations) | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1
Amylase increased (Investigations) | 1
Lipase increased (Investigations) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib (N=129)
Neutropenia (Blood and lymphatic system disorders) | 37
Thrombocytopenia (Blood and lymphatic system disorders) | 25
Anaemia (Blood and lymphatic system disorders) | 36
Diarrhoea (Gastrointestinal disorders) | 63
Nausea (Gastrointestinal disorders) | 38
Vomiting (Gastrointestinal disorders) | 22
Abdominal pain (Gastrointestinal disorders) | 20
Constipation (Gastrointestinal disorders) | 15
Dry mouth (Gastrointestinal disorders) | 9
Stomatitis (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 37
Pyrexia (General disorders) | 32
Oedema peripheral (General disorders) | 22
Asthenia (General disorders) | 15
Chills (General disorders) | 9
Oral Candidiasis (Infections and infestations) | 8
Alanine aminotransferase increased (Investigations) | 17
Aspartate aminotransferase increased (Investigations) | 13
Lipase increased (Investigations) | 12
Weight decreased (Investigations) | 13
Blood alkaline phosphatase increased (Investigations) | 7
Blood creatinine increased (Investigations) | 8
Neutrophil count decreased (Investigations) | 7
Decreased appetite (Metabolism and nutrition disorders) | 19
Hypokalaemia (Metabolism and nutrition disorders) | 18
Dehydration (Metabolism and nutrition disorders) | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8
Headache (Nervous system disorders) | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 35
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 22
Night sweats (Skin and subcutaneous tissue disorders) | 13
Pruritus (Skin and subcutaneous tissue disorders) | 10
Urinary tract infection (Infections and infestations) | 7
Blood lactate dehydrogenase increased (Investigations) | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 7
Dizziness (Nervous system disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-11-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT01882803/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT01882803/SAP_001.pdf